CLINICAL TRIAL: NCT03959579
Title: Long-term Outcomes After Non-invasive Assessment of Acute Cardiac Rejection in Heart Transplantation : the Marie Lannelongue Hospital Experience
Brief Title: The "no Biopsy Approach" for Heart Transplantation Follow-up
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-28
Record Dates: First submitted 2018-05-04; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1st cohort = "derivation cohort":: 1st cohort = "derivation cohort": 1990-1998: cardiac echo + simultaneous systematic endomyocardial biopsy
  Interventions: Diagnostic Test: systematic endomyocardial biopsy.
- 2nd cohort = "validation cohort": 2nd cohort = "validation cohort": 1999-2016: only cardiac echo with same protocol (endomyocardial biopsy only in case of doubt)

INTERVENTIONS:
Diagnostic Test: systematic endomyocardial biopsy. — We sought to compare the long term survival of HTx recipients followed with or without systematic endomyocardial biopsy. Second, the sensibility and specificity of cardiac echo to diagnose acute allograft rejection will be analyzed.
  To show the safety of non-invasively monitoring HTx recipients without systematic endomyocardial biopsy
  Groups: 1st cohort = "derivation cohort":

SUMMARY:
Pathological analysis is the gold standard for diagnosis of acute allograft rejection after heart transplantation (HTx). This method requires repeated endomyocardial biopsies during the first post-operative year. However the sensitivity of endomyocardial biopsy (EMB) is not perfect and can be associated with major complications including fatal tamponade. Moreover, repeated biopsies are associated with reduced quality of life for HTx recipients.

Since almost 20 years, the investigators do not perform routinely EMB for acute rejection screening. Early left ventricular diastolic dysfunction was investigated according to a standardized protocol. The investigators sought to analyze the long-term post-transplant outcomes without systematic EMB. The investigators hypothesize that exclusive echographic screening was not associated with impaired outcomes.

DETAILED DESCRIPTION:
Demographic characteristics of heart transplant recipients and organ donors were prospectively collected in a local database. All HTx successively performed in the Hospital Marie Lannelongue from 1990 to 2016 were included. From 1990 to 1997, both EMB and cardiac echo were routinely performed at each medical follow-up date. After 1997, only cardiac echo was used to detect early acute allograft rejection. The investigators collected the results of all EMB and synchronous cardiac echo in patients transplanted between 1990 and 1997 (group A, validation cohort), and clinical events and long-term survival in patients transplanted from 1998 to 2016 (group B, standardization cohort). For our purpose, the investigators graded the histological patterns of acute cardiac rejection according to the 1990 international classification. Cardiac echo assessment included the isovolumic relaxation time, E-wave velocity and E/A ratio. Impaired left ventricular relaxation was consistent with acute cardiac rejection.

The investigators therefore analyzed the rate of positive and negative EMB during the first post-transplant year and compared these results to the synchronous cardiac echo report in group A. Sensibility and specificity of cardiac echo to detect acute cardiac rejection were calculated. The rate of acute cardiac rejection during the first year was collected in group B and compared to group A. Finally, long-term survival was analyzed according to the Kaplan-Meier approach and compared between group A and B (log-rank test). The investigators hypothesize that the participant will not observe any differences between groups considering the rate of acute cardiac rejection during the first year. In addition, the investigators do not expect to find any significant difference in long-term survival between the two cohorts. These findings may have a major impact on HTx follow-up since systematic EMB could be replaced by a standardized cardiac echo protocol focusing on left ventricular wall relaxation. EMB should therefore only be indicated in case of acute allograft dysfunction without evidence of rejection on conventional cardiac echo.

ELIGIBILITY:
Inclusion Criteria:

* All heart transplant patients, including heart / liver and heart / kidney, and followed at Marie Lannelongue Hospital
* Transplantations carried out between 01/01/1990 and 31/12/2006
* Major and minor patients

Exclusion Criteria:

* Patient with missing test data (cardiac ultrasound or endomyocardial biopsy)
* Patient who did not simultaneously benefit from cardiac ultrasound and endomyocardial biopsy (Delayed period of +/- 1 days)
* Patient who had an endomyocardial biopsy without cardiac ultrasound the day before or the day after endomyocardial biopsy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 269 patients (alive and deceased) patients transplanted between 1990 and 1998 and 1999 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Long-term survival | 15 years
  Survival of patients

SECONDARY OUTCOMES:
Sensitivity | 15 years
  Sensitivity of Cardiac Ultrasound to Diagnose Acute Heart Releases in the 1st Group
Specificity | 15 years
  Specificity of Cardiac Ultrasound to Diagnose Acute Heart Releases in the 1st Group
Positive Predictive Value | 15 years
  Positive Predictive Value of Cardiac Ultrasound to Diagnose Acute Heart Releases in the 1st Group
Negative Predictive Value | 15 years
  Negative Predictive Value of Cardiac Ultrasound to Diagnose Acute Heart Releases in the 1st Group

OTHER OUTCOMES:
Incidence of long-term complications | 15 years
  Incidence of chronic cardiac rejection (coronary disease of the graft), retransplantation rate

CONTACTS AND LOCATIONS:
Overall Officials: Julien Guihaire, MD, PhD, Principal Investigator — Marie Lannelongue Hospital
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No